CLINICAL TRIAL: NCT06421272
Title: APP-based Emotion Recognition Training Improve ASD Social Function
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Weihua Zhao, Associate Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UESTC-neuSCAN-94
Record Dates: First submitted 2024-05-07; First posted 2024-05-20 (Actual); Last update posted 2024-05-20 (Actual); Status verified 2024-05

CONDITIONS: Autism Spectrum Disorder High-Functioning

STUDY DESIGN:
Intervention Model Description: Experimental group (emotion recognition); control group (memory training)
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- APP-based emotion recognition trainning (Experimental): Experimental group: ASD children were asked to do emotion recognition for eight weeks using iPAD. Two 15-minsute sessions each day was required.
  Interventions: Behavioral: APP-based emotion recognition intervention
- APP-based memory training (Active Comparator): Control group: ASD children were asked to do memory training (i.e. 1 back) for eight weeks using iPAD. Two 15-minsute sessions each day was required.
  Interventions: Behavioral: APP-based memory intervention

INTERVENTIONS:
Behavioral: APP-based emotion recognition intervention — ASD children were asked to play emotion recognition-related games for eight weeks using iPAD. Two 15-minsute sessions each day was required.
  Arms: APP-based emotion recognition trainning
Behavioral: APP-based memory intervention — ASD children were asked to play memory-related games for eight weeks using iPAD. Two 15-minsute sessions each day was required.
  Arms: APP-based memory training

SUMMARY:
The main aim of the study is to investigate whether APP-based emotional recognition training improve social function in autistic children.

DETAILED DESCRIPTION:
50 ASD children age ranged from 4-10 years old will be randomly allocated to either app-based emotional recognition training or memory training groups for 2 months. Before and after training, some assessements were measured including Autism Diagnostic Observation Schedule-2, Childhood Autism Rating Scale, Wechsler Intelligence Scale and Psychoeducational Profile-3. Some other questionnaires are also collected including Social Responsibility Scale-2,Repetitive behavior scale-Revised,Caregiver Strains Questionnaire，Social Communication Questionnaire，Social Anxiety Scale for Children，Adaptive behavior assessment Schedule. Four eye-tracking tasks as follows: (1) Dynamic geometrical paired with dynamic child dancing; (2) Static neutral and emotional faces; (3) A dynamic gaze-following task; (4) social interaction behaviors paired with the toys alone; (5) spinning actions conducted via children paired with objects.

ELIGIBILITY:
Inclusion criteria: Clinical diagnosis of Autism Spectrum Disorder and follow these criteria: (1) Age range: 4-10 years old, gender not limited;(2) Ethnicity: Han nationality;(3) Autism Diagnostic Observation Schedule-Second Edition (ADOS-2) Comparison Score greater than or equal to 5 points (Le et al., 2022);(4) Considering that only high-functioning autism individuals can successfully complete the eye-tracking tasks, children with a Wechsler score greater than or equal to 60 points are selected; Exclusion criteria: (1) No neurological complications, such as epilepsy, cerebral palsy, fragile X syndrome, etc.;(2) No prior medical interventions, such as taking antipsychotic drugs, receiving transcranial magnetic stimulation, acupuncture, etc.;(3) No abnormal imaging diagnosis or any brain injury.

Ages: 4 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-05-31 (Estimated); Study Completion 2024-05-31 (Estimated)

PRIMARY OUTCOMES:
ADOS-2 assessment | 1-2 hour
  ADOS-2 assessment
SRS-2 | half an hour
  SRS-2

SECONDARY OUTCOMES:
Visual performance across five tasks based on eye-tracking | half an hour
  Tasked based eye-tracking performance including fixation time, fixation counts

OTHER OUTCOMES:
Other questionnaires and assessment | 1-2 hour
  CARS
Other questionnaires and assessment | 1-2 hour
  PEP-3
Other questionnaires and assessment | 1-2 hour
  RBS-R
Other questionnaires and assessment | 1-2 hour
  SCQ
Other questionnaires and assessment | 1-2 hour
  CSQ

CONTACTS AND LOCATIONS:
Locations (1):
- University of Electronic Science and Technology, Chengdu, Sichuan, China